CLINICAL TRIAL: NCT01732263
Title: A Phase 1, Open-label, Single-dose Study of the Pharmacokinetics, Safety, and Tolerability of SSP-004184 (SPD602) in Subjects With Hepatic Impairment Compared to Matched Healthy Subjects
Brief Title: Study of SSP-004184 (SPD602) in Healthy Adults and Subjects With Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD602-105
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Hepatic Impairment; Healthy
MeSH Terms: interventions — 4,5-dihydro-2-(2-hydroxy-3-(3,6,9-trioxadecyloxy)phenyl)-4-methyl-4-thiazolecarboxylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SSP-004184 (Child-Pugh A Liver Impaired) (Experimental): The Child-Pugh Score is a scoring system used to determine the prognosis with cirrhosis and need for liver transplantation. Scoring is based upon albumin, ascites, total bilirubin, prothrombin time, and encephalopathy. Each category is based on a scoring system of 1-3 with 3 being the worst and a total score range of 5-15. It is broken into categories A (score of 5-6), B (score of 7-9), and C (score of 10-15) with worsening from A to C for prognosis.
  Interventions: Drug: SSP-004184
- SSP-004184 (Child-Pugh B Liver Impaired) (Experimental)
  Interventions: Drug: SSP-004184
- SSP-004184 (Child-Pugh C Liver Impaired) (Experimental)
  Interventions: Drug: SSP-004184
- SSP-004184 (Matched Healthy Subjects) (Experimental)
  Interventions: Drug: SSP-004184

INTERVENTIONS:
Drug: SSP-004184 — All subjects will take a single oral dose of SSP-004184 (SPD602) (50 mg/kg) on Day 1
  Other Names: SPD602, FBS0701

SUMMARY:
The purpose of this study is to evaluate how much of the study drug SSP-004184 (SPD602) is absorbed by the body and how long it takes to be eliminated from the body in healthy subjects and subjects with mild, moderate, and severe hepatic (liver) impairment compared with subjects with healthy normal liver function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years inclusive at the time of consent.
* Willingness to comply with any applicable contraceptive requirements of the protocol and is:
* Male, or
* Non pregnant, non lactating female
* Females must be at least 90 days post partum or nulliparous.

Subjects who do not have hepatic impairment (healthy subjects)

* Normal renal function.

Subjects with hepatic impairment

* Subjects must provide a letter of evaluation from a hepatologist or copy of supporting documents confirming the subject's hepatic impairment (a liver biopsy is preferable but not mandatory).
* Hepatic impairment should be primary and must not be a complication of an underlying primary systemic disease (eg, patients with metastatic cancer and cancer cachexia)
* Documented chronic stable liver impairment

Exclusion Criteria

Subjects who do not have hepatic impairment (healthy subjects)

* A positive HIV antibody screen, Hepatitis B surface antigen, or Hepatitis C virus antibody screen.

Subjects with hepatic impairment

* Presence of a hepatocellular carcinoma, or an acute hepatic disease caused by an infection or drug toxicity.
* Presence of surgically created or transjugular intrahepatic portal systemic shunts.
* A positive HIV antibody screen.
* Renal insufficiency.

All subjects

* Subject has a history of thyroid disorder.
* History of nephrotic syndrome.
* History of alcohol or other substance abuse within the last year.
* A positive screen for alcohol or drugs of abuse.
* Male subjects who consume more than 3 units of alcohol per day. Female subjects who consume more than 2 units of alcohol per day. (1 alcohol unit = 1 beer [12 oz/355 mL] = 1 wine [5 oz/150 mL] = 1 liquor [1.5 oz/40 mL] = 0.75 oz/20 mL alcohol.)
* Caffeine consumption: For healthy subjects: Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches or have a history of caffeine withdrawal headaches. (One caffeine unit is contained in the following items: one 6 oz/180 mL cup of coffee, two 12 oz/355 mL (ie, 24 oz/710 mL cola) cans of cola, one 12 oz/355 mL cup of tea, three 1 oz/28 g chocolate bars (ie, 3 oz/85 g chocolate). Decaffeinated coffee, tea, or cola are not considered to contain caffeine.)
* Donation of blood or blood products within 60 days.
* Substantial changes in eating habits within 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-11-09 (Actual); Primary Completion 2013-04-01 (Actual); Study Completion 2013-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center (OCRC), Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject withdrew from study prior to randomization (n = 43).
Groups:
- Hepatic Impairment; Matched Healthy Subjects: All subjects will take a single oral dose of SSP-004184 (SPD602) (50 mg/kg) on Day 1 (or a revised dose if dose modifications are warranted).
Period: Overall Study
Arm/Group | Hepatic Impairment | Matched Healthy Subjects
Started | 23 | 20
Completed | 23 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hepatic Impairment | Matched Healthy Subjects | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (5.13) | 55.1 (5.51) | 55.7 (5.28)
Age, Customized [Count of Participants; unit: Participants]
  >=65 years | 1 | 0 | 1
  Between 18 and 65 years | 22 | 20 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 19 | 16 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of SSP-004184
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Over 96 hours post-dose
Population: Pharmacokinetic Analysis Set consists of all subjects in the Safety Analysis Set for whom the primary pharmacokinetic data were considered sufficient and interpretable. Safety Analysis Set consists of all enrolled subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Groups:
- SSP-004184 (Child-Pugh A Liver Impaired) 50 mg/kg; SSP-004184 (Child-Pugh B Liver Impaired) 45 mg/kg; SSP-004184 (Child-Pugh B Liver Impaired) 50 mg/kg; SSP-004184 (Child-Pugh C Liver Impaired) 45 mg/kg: The Child-Pugh Score is a scoring system used to determine the prognosis with cirrhosis and need for liver transplantation. Scoring is based upon albumin, ascites, total bilirubin, prothrombin time, and encephalopathy. Each category is based on a scoring system of 1-3 with 3 being the worst and a total score range of 5-15. It is broken into categories A (score of 5-6), B (score of 7-9), and C (score of 10-15) with worsening from A to C for prognosis. All subjects will take a single oral dose of SSP-004184 (SPD602) (50 mg/kg) on Day 1 (or a revised dose if dose modifications are warranted).
- SSP-004184 (Matched Healthy Subjects) 45 mg/kg; SSP-004184 (Matched Healthy Subjects) 50 mg/kg: All subjects will take a single oral dose of SSP-004184 (SPD602) (50 mg/kg) on Day 1 (or a revised dose if dose modifications are warranted).
Arm/Group | SSP-004184 (Child-Pugh A Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 45 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh C Liver Impaired) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 50 mg/kg
Number analyzed (Participants) | 8 | 5 | 3 | 7 | 10 | 10
ng*h/ml | 254327.7 (57645.3) | 443053.5 (157352.1) | 288579.6 (149123.5) | 410414.3 (111201.8) | 209989.8 (83155.2) | 310281.3 (112004.9)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of SSP-004184
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: Over 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SSP-004184 (Child-Pugh A Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 45 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh C Liver Impaired) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 50 mg/kg
Number analyzed (Participants) | 8 | 5 | 3 | 7 | 10 | 10
ng/ml | 98887.5 (29689.1) | 121460.0 (28777.7) | 109166.7 (52920.5) | 123985.0 (34807.1) | 83350.0 (28538.1) | 108890.0 (41016.6)

3. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) for SSP-004184
Description: Tmax is the time after administration of a drug when the maximum plasma concentration in the body is reached.
Time Frame: Over 96 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | SSP-004184 (Child-Pugh A Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 45 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh C Liver Impaired) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 50 mg/kg
Number analyzed (Participants) | 8 | 5 | 3 | 7 | 10 | 10
hours | 1.3 [1.0 to 1.5] | 1.5 [1.0 to 2.5] | 1.5 [1.0 to 1.5] | 1.5 [1.0 to 2.5] | 1.0 [1.0 to 1.5] | 1.0 [1.0 to 2.0]

4. Primary Outcome: Plasma Half-Life (T 1/2) of SSP-004184
Description: The time it takes for the blood plasma concentration of a substance to halve.
Time Frame: Over 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SSP-004184 (Child-Pugh A Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 45 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh C Liver Impaired) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 50 mg/kg
Number analyzed (Participants) | 8 | 5 | 3 | 7 | 10 | 10
hours | 21.91 (17.54) | 11.37 (6.47) | 6.93 (0.94) | 6.79 (3.97) | 12.51 (4.51) | 16.19 (8.62)

5. Primary Outcome: Total Body Clearance (CL/F) of SSP-004184
Description: The rate at which a drug is removed from the body.
Time Frame: Over 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | SSP-004184 (Child-Pugh A Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 45 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh C Liver Impaired) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 50 mg/kg
Number analyzed (Participants) | 8 | 5 | 3 | 7 | 10 | 10
L/h/kg | 0.204 (0.042) | 0.110 (0.035) | 0.198 (0.099) | 0.119 (0.047) | 0.246 (0.097) | 0.182 (0.072)

6. Primary Outcome: Volume of Distribution (Vz/F) of SSP-004184
Description: The distribution of a medication between plasma and the rest of the body.
Time Frame: Over 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | SSP-004184 (Child-Pugh A Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 45 mg/kg | SSP-004184 (Child-Pugh B Liver Impaired) 50 mg/kg | SSP-004184 (Child-Pugh C Liver Impaired) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 45 mg/kg | SSP-004184 (Matched Healthy Subjects) 50 mg/kg
Number analyzed (Participants) | 8 | 5 | 3 | 7 | 10 | 10
L/kg | 6.344 (5.276) | 1.796 (1.210) | 2.043 (1.259) | 1.370 (1.539) | 4.103 (1.420) | 4.086 (2.237)

ADVERSE EVENTS:
Arm/Group | Hepatic Impairment | Matched Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 12/23 | 17/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatic Impairment (N=23) | Matched Healthy Subjects (N=20)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 10 (10) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.